CLINICAL TRIAL: NCT03600480
Title: Investigation of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Dosing of NNC0174-0833 in Combination With Semaglutide in Subjects Being Overweight or With Obesity
Brief Title: A Research Study of How NNC0174-0833 Taken With Semaglutide Works in People Who Are Overweight or Obese
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9838-4395; U1111-1203-6796 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NNC0174-0833+Semaglutide (Experimental): Participants will receive increasing doses of NNC0174-0833 along with semaglutide. The treatment period from first treatment (Day 1) to end of the treatment (Day 141) will be 20 weeks.
  Interventions: Drug: NNC0174-0833; Drug: Semaglutide
- Placebo (NNC0174-0833)+Semaglutide (Active Comparator): Participants will receive placebo (NNC0174-0833) along with semaglutide. The treatment period from first treatment (Day 1) to end of the treatment (Day 141) will be 20 weeks
  Interventions: Drug: Semaglutide; Drug: Placebo (NNC0174-0833)

INTERVENTIONS:
Drug: NNC0174-0833 — Participants will receive increasing dose levels of 0.16 mg, 0.3 mg, 0.6 mg, 1.2 mg, 2.4 mg or 4.5 mg of NNC0174-0833 (subcutaneous [s.c.], in a lifted fold of the abdominal skin) injection once weekly starting with a very low dose and then escalated every 4 weeks to a slightly higher dose each time. Each participant will only be given one dose level.
  Arms: NNC0174-0833+Semaglutide
Drug: Semaglutide — Participants will receive 2.4 mg of semaglutide (s.c., in a lifted fold of the abdominal skin) injection once weekly starting with a very low dose and then escalated every 4 weeks to a slightly higher dose each time.
Drug: Placebo (NNC0174-0833) — Participants will receive once weekly injections of NNC0174-0833 matched placebo.
  Arms: Placebo (NNC0174-0833)+Semaglutide

SUMMARY:
The aim of this study is to find out how NNC0174-0833 taken with semaglutide works in people who are overweight or obese. Both study medicines have been investigated on their own. The study also looks at how the study medicines behave in participant's body and how they are removed from the participant's body. Participants will get 1 of the following 2 treatments - which treatment any participant gets is decided by chance: Semaglutide (a new medicine) and NNC0174-0833 (a potential new medicine), or semaglutide and placebo (a "dummy medicine similar to the study medicine but without active ingredients). Participants will get 2 injections per week for 20 weeks. A study nurse at the clinic will inject the medicine with a needle in a skin fold in the participant's stomach area. The study will last for about 16 months, but duration of participation for any participant will last up to about 7.5 months. Participants will have 28 clinic visits with the study staff and some will be overnight visits. Participants will be asked about their health, medical history and habits including mental health questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of non-childbearing potential, aged 18-55 years (both inclusive) at the time of signing informed consent.
* Body mass index (BMI) between 27.0 and 39.9 kg/sqm (both inclusive) at screening. Overweight should be due to excess adipose tissue, as judged by the investigator.

Exclusion Criteria:

* Any disorder at screening which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol.
* Male subject who is not sexually abstinent or surgically sterilised (vasectomy) and is sexually active with female partner(s) of childbearing potential and is not using a highly effective method of contraception (such as condom with spermicide) combined with a highly effective method of contraception for their non-pregnant female partner(s) (Pearl Index below 1%, such as implants, injectables, oral contraceptives, intrauterine devices, diaphragm or cervical cap+spermicide), and/or intend to donate sperm in the period from screening until 3 months following administration of the last dose of investigational medical product.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From first administration of NNC0174-0833 (Day 1) to completion of the post-treatment follow-up (Day 176)
  Count of events

SECONDARY OUTCOMES:
AUC0-168h,AM833,SS: the area under the NNC0174-0833 plasma concentration-time curve from 0 to 168 hours at steady state | From last dose (Day 134) until end of treatment (Day 141)
  Measured in nmol*h/L
Cmax,AM833,SS: the maximum concentration of NNC0174-0833 in plasma at steady state | From last dose (Day 134) until end of treatment (Day 141)
  Measured in nmol/L
AUC0-168h,sema,SS: the area under the semaglutide plasma concentration-time curve from 0 to 168 hours at steady state | From last dose (Day 134) until end of treatment (Day 141)
  Measured in nmol*h/L
Cmax,sema,SS: the maximum concentration of semaglutide in plasma at steady state | From last dose (Day 134) until end of treatment (Day 141)
  Measured in nmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure 1452, Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisktrials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Enebo LB, Berthelsen KK, Kankam M, Lund MT, Rubino DM, Satylganova A, Lau DCW. Safety, tolerability, pharmacokinetics, and pharmacodynamics of concomitant administration of multiple doses of cagrilintide with semaglutide 2.4 mg for weight management: a randomised, controlled, phase 1b trial. Lancet. 2021 May 8;397(10286):1736-1748. doi: 10.1016/S0140-6736(21)00845-X. Epub 2021 Apr 22. PMID 33894838